CLINICAL TRIAL: NCT02390804
Title: Postoperative Pain After Total Laparoscopic Hysterectomy: a Comparison of Transumbilical Single-port Access and Conventional Three-port Laparoscopic Surgery
Brief Title: Postoperative Pain After Total Laparoscopic Hysterectomy: a Comparison of Single-port and Three-port Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong Seok Lee, associated professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DC14EISI0026
Record Dates: First submitted 2015-03-02; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Uterine Disease; Postoperative Pain
Keywords: postoperative pain; hysterectomy; single-port access laparoscopy; multi-port access laparoscopy; TLH
MeSH Terms: conditions — Uterine Diseases; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single-port laparoscopic hysterectomy (Experimental): total laparoscopic hysterectomy via transumbilical single port
  Interventions: Device: single-port laparoscopic hysterectomy(single port trochar)
- multi-port laparoscopic hysterectomy (Active Comparator): total laparoscopic hysterectomy via multi-port (3 port)
  Interventions: Device: multi-port laparoscopic hysterectomy(multi port trochar)

INTERVENTIONS:
Device: single-port laparoscopic hysterectomy(single port trochar) — perform laparoscopic hysterectomy via single-port access
  Arms: single-port laparoscopic hysterectomy
Device: multi-port laparoscopic hysterectomy(multi port trochar) — perform laparoscopic hysterectomy via multi-port access
  Arms: multi-port laparoscopic hysterectomy

SUMMARY:
The objective of this study is to compare postoperative pain between single-port access total laparoscopic hysterectomy (SPA-TLH) using a transumbilical single-port system and conventional multi (three)-port access total laparoscopic hysterectomy (MPA-TLH). A prospective study was conducted on women who underwent SPA-TLH and MPA-TLH for benign gynecologic diseases from March 2014 through January 2015. The study enrolled 60 patients and postoperative pain and operative outcomes were examined.

DETAILED DESCRIPTION:
The randomization code was inserted into numbered and sealed envelopes. A single envelope was opened when the patient was arrived in operating room. All patients gave their informed consent for the study and underwent hysterectomy for benign diseases. After surgery, in all patients, three sticking plasters were applied by the same manner with three port surgery group therefore not only patients but also anesthesiology staff who measure the pain score could not know the type of surgery until data collection was finished. Pain was assessed according to the visual analog scale (VAS) (0 = no pain; 10 = worst pain imaginable). Patients were asked to evaluate the maximal degree of pain. Pain scores were recorded at least at 30 minutes, 1, 12, 24 and 48 hours after surgery. Postoperative pain was measured by two independent anesthesiology staff members for cross-checking. In order to compare the intensity of postoperative pain accurately, all the participants had anesthesia in the same way and postoperative pain was managed by fentanyl-based intravenous patient-controlled analgesia pump (IV-PCA, Baxter healthcare Corporation, U.S.A: bolus dose 0.12mg/kg of fentanyl, lockout interval of 5 min, basal infusion 0.02ml/kg) with the same regimen on both groups. A patient was instructed to press the IV-PCA bolus button when the VAS was 3 or higher. A patient under IV-PCA whose VAS was over 5 received 50mg of Tridol injection intravenously. IV-PCA was removed 48 hours after surgery unless a patient specially asked it. Then, using log data downloaded by a program, we analyzed the number of IV-PCA bolus requests by time interval, total amount of fentanyl consumption, and the number of additional Tridol administration and injection time.

ELIGIBILITY:
Incluson Criteria

1. Subject has benign uterine disease
2. Subject needs total hysterectomy.
3. Subject has appropriate medical status for laparoscopic surgery (American Society of Anesthesiologists Physical Status classification system 1-3).

Exclusion Criteria:

1. suspicion of malignancy
2. the need for simultaneous interventions such as prolapse repair
3. uterine size greater than 18 weeks of gestation
4. ongoing peritoneal dialysis
5. diseases associated with abdominal pain such as pancreatitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain (Pain scores) intensity measure | 2 days
  self reported pain intensity measure for 2 days after surgery

SECONDARY OUTCOMES:
Number of Participants with Adverse events | up to 24 weeks
  perioperative adverse event including bowel, bladder injury and severe hemorrahge

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Hyun Chung, MD, Study Director — The Catholic University of Korea

REFERENCES:
- [Background] Lee YY, Kim TJ, Kim CJ, Kang H, Choi CH, Lee JW, Kim BG, Lee JH, Bae DS. Single-port access laparoscopic-assisted vaginal hysterectomy: a novel method with a wound retractor and a glove. J Minim Invasive Gynecol. 2009 Jul-Aug;16(4):450-3. doi: 10.1016/j.jmig.2009.03.022. Epub 2009 May 31. PMID 19487164
- [Background] Jung YW, Kim YT, Lee DW, Hwang YI, Nam EJ, Kim JH, Kim SW. The feasibility of scarless single-port transumbilical total laparoscopic hysterectomy: initial clinical experience. Surg Endosc. 2010 Jul;24(7):1686-92. doi: 10.1007/s00464-009-0830-7. Epub 2009 Dec 25. PMID 20035346
- [Background] Ng PC. Re: Surg Endosc (2009) 23:1142-1145, DOI:10.1007/s00464-009-0382-x (published online 5 March 2009). Erica P. Podolsky, Steven J. Rottman, Paul G. Curcillo II. Single Port Access (SPA) gastrostomy tube in patients unable to receive percutaneous endoscopic gastrostomy placement. Surg Endosc. 2010 Apr;24(4):970. doi: 10.1007/s00464-009-0705-y. No abstract available. PMID 19789919
- [Background] Fagotti A, Bottoni C, Vizzielli G, Gueli Alletti S, Scambia G, Marana E, Fanfani F. Postoperative pain after conventional laparoscopy and laparoendoscopic single site surgery (LESS) for benign adnexal disease: a randomized trial. Fertil Steril. 2011 Jul;96(1):255-259.e2. doi: 10.1016/j.fertnstert.2011.04.006. Epub 2011 May 11. PMID 21565338
- [Background] Song T, Kim ML, Jung YW, Yoon BS, Joo WD, Seong SJ. Laparoendoscopic single-site versus conventional laparoscopic gynecologic surgery: a metaanalysis of randomized controlled trials. Am J Obstet Gynecol. 2013 Oct;209(4):317.e1-9. doi: 10.1016/j.ajog.2013.07.004. Epub 2013 Jul 13. PMID 23860211
- [Background] Eom JM, Choi JS, Choi WJ, Kim YH, Lee JH. Does single-port laparoscopic surgery reduce postoperative pain in women with benign gynecologic disease? J Laparoendosc Adv Surg Tech A. 2013 Dec;23(12):999-1005. doi: 10.1089/lap.2013.0184. Epub 2013 Oct 1. PMID 24083850